CLINICAL TRIAL: NCT06991920
Title: Immune-targeted Combination With Acute Lymphoblastic Leukemia-like Chemotherapy for Adult of Acute Leukemia of Ambiguous Lineage: A Prospective, Single-arm, Multicenter Clinical Study
Brief Title: Immune-targeted Combination With Chemotherapy for Acute Leukemia of Ambiguous Lineage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024114
Record Dates: First submitted 2025-03-17; First posted 2025-05-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-03

CONDITIONS: Adult ALL; MPAL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systematic treatment strategy (Experimental): Integrate Blinatumomab, ALL-like chemotherapy, Venetoclax and TKI drugs into the systemic treatment plan
  Interventions: Drug: Blinatumomab; Drug: Venetoclax

INTERVENTIONS:
Drug: Blinatumomab — CD19-positive, Ph+ patients with favorable financial status may receive VP + TKI + blinatumomab therapy；CD19-positive, Ph- patients with favorable financial status may receive VCP + blinatumomab therapy.
Drug: Venetoclax — CD19-positive, Ph+ patients with poor financial status may receive VP + TKI + VEN therapy；CD19-negative or CD19-positive, Ph- patients ineligible for blinatumomab may receive VPCLP + VEN therapy.

SUMMARY:
Acute leukemia of ambiguous lineage (ALAL), which refers to acute leukemia without definite evidence indicating cell differentiation along a specific lineage, mainly encompasses two major categories: acute undifferentiated leukemia (AUL) lacking the expression of lineage-specific antigens and mixed phenotype acute leukemia (MPAL) expressing antigens of two or more lineages. Despite certain advancements in basic research on ALAL, there is currently no unified treatment protocol for this disease. The majority of clinical studies are based on retrospective data, lacking prospective cohort studies. In terms of the overall treatment strategy, given the low chemotherapy remission rate, frequent relapses, and poor prognosis of ALAL, it should be treated as high-risk acute leukemia. Patients achieving complete remission should undergo allogeneic hematopoietic stem cell transplantation as soon as possible if conditions permit. Regarding chemotherapy regimens, the current main regimens utilized in clinical practice include ALL-like regimens, AML-like regimens, and hybrid therapies that incorporate both lymphoid and myeloid lineages. Based on existing research, international consensus guidelines recommend ALL-like regimens as the preferred induction treatment option for ALAL patients. In recent years, novel immunotherapy antibody drugs, such as Blinatumomab (a CD19-targeted drug), have achieved remarkable success in the treatment of B-ALL. However, for CD19+ ALAL, there is a lack of effective data regarding whether the first-line application of immunotherapy can further enhance therapeutic efficacy. Simultaneously, the novel small molecule drug venetoclax has demonstrated favorable therapeutic effects on various hematological malignancies. To enhance the overall therapeutic efficacy of adult ALAL in China, based on the above research, we have formulated a comprehensive treatment plan for adult ALAL, integrating Blinatumomab, ALL-like chemotherapy, venetoclax, and TKI drugs into the systemic treatment regimen, and exploring the safety and efficacy of this regimen in the treatment of adult ALAL.

ELIGIBILITY:
Inclusion Criteria:

* A series of acute leukemia of unknown origin diagnosed in accordance with the 5th edition of the WHO or ICC classification standards.
* Age ≥ 14 years old, regardless of gender.
* The ECOG performance status score is ≤ 2.
* Conform to the following organ functional status: total bilirubin < 1.5×ULN, AST and ALT ≤ 2.5×ULN; blood Cr < 1.5×ULN; myocardial enzymes < 2×ULN; serum amylase ≤ 1.5×ULN; echocardiography indicates that the left ventricular ejection fraction (LEF) > 50%. (In the case of patients without a previous history of liver or kidney basic disease, if liver and kidney function abnormalities exceed the aforementioned inclusion criteria and the researcher determines that the liver and kidney function abnormalities are caused by acute leukemia itself, they may be included in the group at the researcher's discretion).
* Understand and sign the informed consent form and agree to abide by the research requirements.

Exclusion Criteria:

* Concurrent with other serious and/or uncontrollable underlying diseases: accompanied by other malignant diseases requiring treatment, acute or chronic hepatitis, severe pancreatic or kidney diseases; other serious and/or life-threatening underlying diseases.
* Pregnant or lactating women.
* Positive for anti-HIV test.
* Mental disorders that may prevent the subject from completing the treatment or giving informed consent.
* The investigator deems the subject unsuitable for inclusion.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | up to 2 years
  Used to evaluate all patients who enter clinical trials. From the date of entry into the trial until the date of patient death (including any cause) or last survival follow-up.

SECONDARY OUTCOMES:
Complete remission (CR) rate or complete remission with partial hematologic recovery (CRh) rate or complete remission with incomplete hematologic recovery (CRi) rate | Six weeks after induction therapy
  Proportion of patients with CR, CRh or Cri
Flow cytometry for minimal residual disease（FCM-MRD） negativity rate at 3 months post-therapy | 3 months after therapy
  FCM-MRD is a method that detects residual trace leukemia or lymphoma cells in patients' bodies after treatment
Relapse free survival(RFS) | up to 2 years after the date of the last enrolled participants
  The interval from CR to the date of relapse, or the date of death, or the date of last follow-up, whichever occurred first. This outcome analyzes patients achieved CR in two courses of induction therapy.
Event-free survival (EFS) | up to 2 years after the date of the last enrolled participants
  The interval from the date of enrollment to the date of failed to achieve complete remission, the date of relapse, or the date of death, whichever occurred first.
Disease-free Survival (DFS) | up to 2 years after the date of the last enrolled participants
  From CR1 to relapse, death from any cause or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wei, MD, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College